CLINICAL TRIAL: NCT04626102
Title: Healthy Eating Attitudes and Behaviours Group Program: A Randomised Controlled Feasibility Study
Brief Title: Healthy Eating Attitudes and Behaviours Group Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Arel University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Başak İnce, Research Assistant, Istanbul Arel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IstanbulArelU
Record Dates: First submitted 2020-10-30; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Eating Disorders; Body Image Disturbance
Keywords: eating disorders; prevention; university students; cognitive behavioural
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Eligible participants were randomly assigned to 6-session Healthy Eating Attitudes and Behaviours Group Program (experimental group condition), single session Eating Disorders and Body Dissatisfaction: A Group Work (active control group condition) or wait-list control group condition.
Who Masked: Outcomes Assessor
Masking Description: Participants were informed that they are invited to attend a group intervention aiming to improve healthy eating attitudes and behaviours. However, they were not informed that they were invited because they had higher levels of disordered eating attitudes and behaviours than the others who were not invited. Also, they did not know that the real aim was to prevent development of eating disorders.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enrollment (No Intervention): Participants were recruited by using a convenience sampling method. Potential participants were reached through lecturers and professors who are teaching classes at different universities in Istanbul, Turkey.
  Participants were asked to fill out a questionnaire package covering Demographic Information Form, Eating Disorders Examination Questionnaire (EDEQ), Eating Attitudes Test - 40 (EAT-40), Body Image Satisfaction Questionnaire (BISQ), and Sociocultural Attitudes towards Appearance Questionnaire-4-Revised (SATAQ-4R). Filling out the questionnaire package took approximately 25-minutes.
- Intervention Period (Experimental): Participants were randomly assigned to one of these conditions:
  Experimental condition: Healthy Eating Attitudes and Behaviours Group Program - 6 weekly sessions, each session was about 45-minutes to 60-minutes
  Active control condition: Eating Disorders and Body Dissatisfaction: A Group Work - single session about 1.5 hours to 2 hours
  Wait-list control condition: Participants in this condition were informed that they will be asked to fill out questionnaires that sent to them, and at the end of 6 months, they will be invited to participate in Healthy Eating Attitudes and Behaviours Group Program.
  Interventions: Behavioral: Healthy Eating Attitudes and Behaviours Group Program (Experimental Group Condition); Behavioral: Eating Disorders and Body Dissatisfaction: A Group Work (Active Control Group Condition)

INTERVENTIONS:
Behavioral: Healthy Eating Attitudes and Behaviours Group Program (Experimental Group Condition) — The program has been developed by Clinical Psychologist Başak İnce and Psychiatrist Prof. Dr Başak Yücel. The session topics and contents of this program were based on the Fairburn (2008)'s book titled Cognitive- Behavior Treatment and Eating Disorders and 10-week online version of StudentBodies program designed by Saekow and her colleagues (2015). Program protocol was written based on Fairburn (2008)'s book titled Cognitive- Behavior Treatment and Eating Disorders and Fursland and her colleagues (2007)'s book titled Overcoming Disordered Eating.
  This program aimed to inform participants about the causes and consequences of eating disorders, teach cognitive and behavioural techniques to change their unhealthy eating attitudes and behaviours, and provide support during their attitudinal and behavioural changes. Each week, participants were asked to complete homework activities which were related to topics covered in each session.
  Arms: Intervention Period
Behavioral: Eating Disorders and Body Dissatisfaction: A Group Work (Active Control Group Condition) — This single-session group program was designed as an active control group for the purpose of this study. The content of the program was prepared based on Stice and his colleagues (2013)'s four - sessions Body Project eating disorders prevention program. This single-session program aimed to inform participants about causes and consequences of eating disorders, and discuss "thin ideal" messages created by media and the negative impact of these messages on women's body images, and address possible ways of countering these messages. Detailed information regarding the covered topics and video presentations in the group session is provided below.
  Arms: Intervention Period

SUMMARY:
Eating disorders (ED) are serious mental health illnesses interfering psychological, physical and social well-being. Besides the severity of ED, most of the individuals presenting symptoms are either not detected or treated. Among ones undergoing treatment, full recovery and remission are also not very likely. Given many negative consequences of ED and personal, sociocultural and financial barriers for ED treatment and low rates of full recovery, any intervention for preventing the development and/or chronicization of ED would be a useful step for the improvement of public health.

Literature has established that Turkish people represent unhealthy eating attitudes and behaviours as similar to Western societies. Evidence shows that the prevalence of disordered eating attitudes and behaviours in Turkey changed between 2.2% to 12.8%. Prevalence of ED particularly among university students and these problems are also likely to negatively influence students' psychological, social and physical well-being, relationships with pairs, educational attainment and academic success. However, awareness regarding ED, help-seeking and receiving treatment appears to be less likely.

Since there is no ED prevention program available for university students in Turkey, it was aimed to develop a Cognitive Behaviour Therapy oriented 6 session ED prevention program (Healthy Eating Attitudes and Behaviours Group Program) for female university students presenting a high risk for ED. A further aim was to examine feasibility, acceptability and efficacy of this program.

Evidence-based clinical guidelines for ED have indicated that CBT is consistently recommended for all subtypes of ED, and CBT oriented prevention programs have been shown to result in a better outcome for university students. Therefore, it was expected that university students who participated in 6 session Healthy Eating Attitudes and Behaviours Group Program would present significantly greater reductions in ED related psychopathology, body dissatisfaction, emotion regulation difficulties and internalization and pressure of sociocultural attitudes towards appearance compared to participants in active control group condition (single session Eating Disorders and Body Dissatisfaction: A Group Work) and wait-list control condition. Also, it was expected that the level of acceptability and feasibility of 6 session Healthy Eating Attitudes and Behaviours Group Program would be good.

ELIGIBILITY:
Inclusion Criteria:

* having a score of EDEQ-Total or EAT - 40 higher than the mean average of female participants in a study conducted among university students in Turkey before
* giving consent during the above-mentioned study for getting an invitation for participating in a study in which a group program for promoting healthy eating attitudes and behaviours.

Exclusion Criteria:

* current or history of eating disorders diagnosis,
* current substance abuse problem and/or current or past history of psychotic disorders.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
The Eating Disorders Examination Questionnaire | Arm1: Enrollment; Arm2: Baseline(first day of the group intervention), post-treatment (6 weeks after baseline measurement), 1 month follow up (10 weeks after te baseline measurement)
  This questionnaire was used for measuring restraint eating, shape concern, weight concern, eating concern and general eating disorders related psychopathology. There are four subscales named Restraint, Eating Concern, Shape Concern and Weight Concern, and a total score. The minimum score for this scale is 0, while the maximum score is 6. Higher scores indicate greater levels of disordered eating attitudes and behaviours. This questionnaire was used to assess the level of change from baseline to post-treatment and from baseline to 1 month follow up.
The Body Shape Questionnaire | Arm2: Baseline(first day of the group intervention), post-treatment (6 weeks after baseline measurement), 1 month follow up (10 weeks after te baseline measurement)
  This questionnaire was used for measuring preoccupation with body weight and shape. Scores can range from 34 (minimum) to 204 (maximum). Higher scores indicate greater levels of body dissatisfaction. This questionnaire was used to assess the level of change from baseline to post-treatment and from baseline to 1 month follow up.

SECONDARY OUTCOMES:
The Difficulties in Emotion Regulation Scale -16 | Arm2: Baseline(first day of the group intervention), post-treatment (6 weeks after baseline measurement), 1 month follow up (10 weeks after te baseline measurement)
  This questionnaire was used for measuring different aspects of emotion regulation difficulties. The minimum score for this scale is 0, while the maximum score is 64. Higher scores indicate greater levels of difficulty in emotion regulation. This questionnaire was used to assess the level of change from baseline to post-treatment and from baseline to 1 month follow up.
The Sociocultural Attitudes towards Appearance Questionnaire-4-Revised | Arm2: Baseline(first day of the group intervention), post-treatment (6 weeks after baseline measurement), 1 month follow up (10 weeks after te baseline measurement)
  This questionnaire was used for measuring the influence of societal and interpersonal influences on body image and disturbances in eating behaviour. There are 7 subscales of this questionnaires: (1) Internalization: Thin/Low Body Fat, (2) Internalization: Muscular, (3) Internalization: General Attractiveness, (4) Pressures: Family, (5) Pressures: Media, (6) Pressures: Peers, and (7) Pressures: Significant Others. For each subscale, scores can range from 1 (minimum) to 5 (maximum). Higher scores indicate greater levels of internalization or pressures.
  This questionnaire was used to assess the level of change from baseline to post-treatment and from baseline to 1 month follow up.

OTHER OUTCOMES:
The Eating Attitudes Test - 40 | Arm1: Enrollment
  This questionnaire was used to measure disordered eating attitudes and behaviours. Score of 30 and greater indicates greater disordered eating attitudes.
The Group Feedback Form | Arm 2: Post-treatment (6 weeks after baseline measurement)
  feedback form was designed in order to gather information about the satisfaction with the aspects of the group program (e.g., structure, helpfulness, content of the program, the quality/features of the group therapist).

CONTACTS AND LOCATIONS:
Overall Officials: Başak Yücel, MD, Study Director — Professor
Locations (1):
- Istanbul Arel University, Istanbul, Sefaköy-Küçükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fairburn CG. Cognitive behavior therapy and eating disorders: Guilford Press. 2008. 323 p.
- [Background] Kugu N, Akyuz G, Dogan O, Ersan E, Izgic F. The prevalence of eating disorders among university students and the relationship with some individual characteristics. Aust N Z J Psychiatry. 2006 Feb;40(2):129-35. doi: 10.1080/j.1440-1614.2006.01759.x. PMID 16476130
- [Background] Saekow J, Jones M, Gibbs E, Jacobi C, Fitzsimmons-Craft EE, Wilfley D, & Barr Taylor C. StudentBodies-eating disorders: A randomized controlled trial of a coached online intervention for subclinical eating disorders. Internet Interventions. 2015; 2(4): 419-428. doi:https://doi.org/10.1016/j.invent.2015.10.004
- [Background] Stice E, Butryn ML, Rohde P, Shaw H, Marti CN. An effectiveness trial of a new enhanced dissonance eating disorder prevention program among female college students. Behav Res Ther. 2013 Dec;51(12):862-71. doi: 10.1016/j.brat.2013.10.003. Epub 2013 Oct 19. PMID 24189570
- [Background] Taylor CB, Bryson S, Luce KH, Cunning D, Doyle AC, Abascal LB, Rockwell R, Dev P, Winzelberg AJ, Wilfley DE. Prevention of eating disorders in at-risk college-age women. Arch Gen Psychiatry. 2006 Aug;63(8):881-8. doi: 10.1001/archpsyc.63.8.881. PMID 16894064
- [Background] Watson HJ, Joyce T, French E, Willan V, Kane RT, Tanner-Smith EE, McCormack J, Dawkins H, Hoiles KJ, Egan SJ. Prevention of eating disorders: A systematic review of randomized, controlled trials. Int J Eat Disord. 2016 Sep;49(9):833-62. doi: 10.1002/eat.22577. Epub 2016 Jul 18. PMID 27425572
- [Background] Yucel B, Polat A, Ikiz T, Dusgor BP, Elif Yavuz A, Sertel Berk O. The Turkish version of the eating disorder examination questionnaire: reliability and validity in adolescents. Eur Eat Disord Rev. 2011 Nov-Dec;19(6):509-11. doi: 10.1002/erv.1104. Epub 2011 Mar 13. PMID 21400637
- [Background] White S, Reynolds-Malear JB, Cordero E. Disordered eating and the use of unhealthy weight control methods in college students: 1995, 2002, and 2008. Eat Disord. 2011 Jul-Aug;19(4):323-34. doi: 10.1080/10640266.2011.584805. PMID 22352972
- [Background] Vardar E, Erzengin M. The prevalence of eating disorders (EDs) and comorbid psychiatric disorders in adolescents: a two-stage community-based study. Turk Psikiyatri Derg. 2011 Winter;22(4):205-12. PMID 22143945
- [Background] Stice E, Shaw H, Marti CN. A meta-analytic review of eating disorder prevention programs: encouraging findings. Annu Rev Clin Psychol. 2007;3:207-31. doi: 10.1146/annurev.clinpsy.3.022806.091447. PMID 17716054
- [Background] Schaefer LM, Harriger JA, Heinberg LJ, Soderberg T, Kevin Thompson J. Development and validation of the sociocultural attitudes towards appearance questionnaire-4-revised (SATAQ-4R). Int J Eat Disord. 2017 Feb;50(2):104-117. doi: 10.1002/eat.22590. Epub 2016 Aug 19. PMID 27539814
- [Background] Linardon J, Fairburn CG, Fitzsimmons-Craft EE, Wilfley DE, Brennan L. The empirical status of the third-wave behaviour therapies for the treatment of eating disorders: A systematic review. Clin Psychol Rev. 2017 Dec;58:125-140. doi: 10.1016/j.cpr.2017.10.005. Epub 2017 Oct 23. PMID 29089145
- [Background] Hay P. Current approach to eating disorders: a clinical update. Intern Med J. 2020 Jan;50(1):24-29. doi: 10.1111/imj.14691. PMID 31943622
- [Background] Griffiths S, Rossell SL, Mitchison D, Murray SB, Mond JM. Pathways into treatment for eating disorders: A quantitative examination of treatment barriers and treatment attitudes. Eat Disord. 2018 Nov-Dec;26(6):556-574. doi: 10.1080/10640266.2018.1518086. Epub 2018 Sep 17. PMID 30222057
- [Background] Gratz KL, & Roemer L. Multidimensional Assessment of Emotion Regulation and Dysregulation: Development, Factor Structure, and Initial Validation of the Difficulties in Emotion Regulation Scale. Journal of Psychopathology and Behavioral Assessment. 2004; 26(1): 41-54. doi:10.1023/b:Joba.0000007455.08539.94
- [Background] Garner DM, Garfinkel PE. The Eating Attitudes Test: an index of the symptoms of anorexia nervosa. Psychol Med. 1979 May;9(2):273-9. doi: 10.1017/s0033291700030762. PMID 472072
- [Background] Fursland A, Byrne S, & Nathan P. Overcoming disordered eating. Centre for Clinical Interventions. 2007
- [Background] Fairburn CG, Cooper Z, Shafran R. Cognitive behaviour therapy for eating disorders: a "transdiagnostic" theory and treatment. Behav Res Ther. 2003 May;41(5):509-28. doi: 10.1016/s0005-7967(02)00088-8. PMID 12711261
- [Background] Fairburn CG, Beglin SJ. Assessment of eating disorders: interview or self-report questionnaire? Int J Eat Disord. 1994 Dec;16(4):363-70. PMID 7866415
- [Background] Evans EJ, Hay PJ, Mond J, Paxton SJ, Quirk F, Rodgers B, Jhajj AK, Sawoniewska MA. Barriers to help-seeking in young women with eating disorders: a qualitative exploration in a longitudinal community survey. Eat Disord. 2011 May-Jun;19(3):270-85. doi: 10.1080/10640266.2011.566152. PMID 21516551
- [Background] Evans C, Dolan B. Body Shape Questionnaire: derivation of shortened "alternate forms". Int J Eat Disord. 1993 Apr;13(3):315-21. doi: 10.1002/1098-108x(199304)13:33.0.co;2-3. PMID 8477304
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. Pilot Feasibility Stud. 2016 Oct 21;2:64. doi: 10.1186/s40814-016-0105-8. eCollection 2016. PMID 27965879
- [Background] Cok F. Body image satisfaction in Turkish adolescents. Adolescence. 1990 Summer;25(98):409-13. PMID 2375266
- [Background] Cihan B, Bozo O, Schaefer LM, Thompson JK. Psychometric properties of the Sociocultural Attitudes Towards Appearance Questionnaire-4-Revised (SATAQ-4R) in Turkish women. Eat Behav. 2016 Apr;21:168-71. doi: 10.1016/j.eatbeh.2016.03.003. Epub 2016 Mar 4. PMID 26970730
- [Background] Ciao AC, Loth K, Neumark-Sztainer D. Preventing eating disorder pathology: common and unique features of successful eating disorders prevention programs. Curr Psychiatry Rep. 2014 Jul;16(7):453. doi: 10.1007/s11920-014-0453-0. PMID 24821099
- [Background] Celikel FC, Cumurcu BE, Koc M, Etikan I, Yucel B. Psychologic correlates of eating attitudes in Turkish female college students. Compr Psychiatry. 2008 Mar-Apr;49(2):188-94. doi: 10.1016/j.comppsych.2007.09.003. Epub 2007 Dec 21. PMID 18243893
- [Background] Brockmeyer T, Skunde M, Wu M, Bresslein E, Rudofsky G, Herzog W, Friederich HC. Difficulties in emotion regulation across the spectrum of eating disorders. Compr Psychiatry. 2014 Apr;55(3):565-71. doi: 10.1016/j.comppsych.2013.12.001. Epub 2013 Dec 7. PMID 24411653
- [Background] Bjureberg J, Ljotsson B, Tull MT, Hedman E, Sahlin H, Lundh LG, Bjarehed J, DiLillo D, Messman-Moore T, Gumpert CH, Gratz KL. Development and Validation of a Brief Version of the Difficulties in Emotion Regulation Scale: The DERS-16. J Psychopathol Behav Assess. 2016 Jun;38(2):284-296. doi: 10.1007/s10862-015-9514-x. Epub 2015 Sep 14. PMID 27239096